CLINICAL TRIAL: NCT03552432
Title: The Efficacy of Alirocumab for Thin-cap fIbroatheroma in Patients With Coronary Artery Disease Estimated by Optical Coherence Tomography: Single Center, Randomized, Open-label, Trial
Brief Title: The Efficacy of Alirocumab for Thin-cap fIbroatheroma in Patients With Coronary Artery Disease Estimated by Optical Coherence Tomography
Acronym: ALTAIR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kobe University (Industry)
Responsible Party: Principal Investigator, Hiromasa Otake, Senior Lecturer, Kobe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KobeU-290017
Record Dates: First submitted 2018-05-07; First posted 2018-06-11 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Coronary Artery Disease; Thin-cap fIbroatheroma
Keywords: alirocumab; Thin-cap fIbroatheroma (TCFA); vulnerable plaque; Optical Coherence Tomography (OCT)
MeSH Terms: conditions — Coronary Artery Disease | interventions — alirocumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alirocumab therapy group (Experimental): start with alirocumab 75mg per 2weeks and rosuvastatin 10mg per day
  Interventions: Drug: Alirocumab
- standard statin therapy group (No Intervention): start with only rosuvastatin 10mg per day

INTERVENTIONS:
Drug: Alirocumab — the administration of Alirocumab by Subcutaneous injection 75mg every 2 weeks plus Rosuvastatin10mg/daily by oral for 9 months
  Arms: Alirocumab therapy group

SUMMARY:
the purpose of this study is to show that alirocumab with statin therapy have a s tronger stabilizing effect on vulnerable plaque in coronary artery disease than statin alone administration

DETAILED DESCRIPTION:
The investigators investigate to evaluate the efficacy of alirocumab for vulnerable plaque. The investigators enrolled the patient with standard statin therapy who were detected vulnerable plaque by optical coherence tomography, and categorized into two group; the patients with alirocumab and rosuvastatin were categorized alirocumab therapy group, and the patients with rosuvastatin alone were categorized standard statin therapy group. The investigators compare these two group for outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent PCI for ACS or stable coronary heart disease
2. Patients with LDL-C ≥70 mg/dL under daily 10mg rosuvastatin
3. Patients who have been had TCFA detected by OCT
4. Patients aged ≥20 years old at PCI
5. Patients who agree to be enrolled in the trial giving signed written informed consent

Exclusion Criteria:

1. Patients who have been treated previously with at least one dose of any anti-PCSK9 monoclonal antibody
2. Patients had uncontrolled hypertension (systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg) between the time of PCI and randomization visit
3. Known hypersensitivity to alirocumab or rosuvastatin
4. All contraindications to alirocumab and/or rosuvastatin as displayed in the respective national product labeling for these treatments
5. Known history of hemorrhagic stroke
6. Currently under treatment for cancer
7. Patients on lipoprotein apheresis
8. Patients with severe liver or renal dysfunction
9. Pregnant or breast-feeding women
10. Considered by the investigator as inappropriate for this study for any reason

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-08-23 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
the change in fibrous cap thickness | 9 month
  the absolute change in minimum fibrous-cap thickness between baseline and 36-week follow-up

SECONDARY OUTCOMES:
the change in fibrous cap thickness | 9 month
  the percent change in minimum fibrous-cap thickness between baseline and 36-week follow-up
the change in lipid index | 9 month
  absolute change in lipid index between baseline and 36-week follow-up
the change in lipid index | 9 month
  percentage change in lipid index between baseline and 36-week follow-up
the change in lipid length, | 9 month
  absolute change in lipid core length between baseline and 36-week follow-up
the change in lipid length, | 9 month
  percentage change in lipid core length between baseline and 36-week follow-up
the change in mean lipid arc | 9 month
  absolute change in mean lipid arc between baseline and 36-week follow-up
the change in mean lipid arc | 9 month
  percentage change in mean lipid arc between baseline and 36-week follow-up
the change in max lipid arc | 9 month
  absolute change in max lipid arc between baseline and 36-week follow-up
the change in max lipid arc | 9 month
  percent change in max lipid arc between baseline and 36-week follow-up
the change in macrophage grade | 9 month
  absolute change in summation of macrophage grade between baseline and 36-week follow-up.
  macrophage grade defined as an OCT macrophage grading system to semiquantify the bright spots based on axial and circumferential distribution, as follows: grade 0, no macrophage; grade 1, localized macrophage accumulation; grade 2, clustered accumulation <1 quadrant; grade 3, clustered accumulation >1 quadrant and ≦3 quadrants; and grade 4, clustered accumulation ≧3
the change in macrophage grade | 9 month
  percentage change in summation of macrophage grade between baseline and 36-week follow-up.
  macrophage grade defined as an OCT macrophage grading system to semiquantify the bright spots based on axial and circumferential distribution, as follows: grade 0, no macrophage; grade 1, localized macrophage accumulation; grade 2, clustered accumulation <1 quadrant; grade 3, clustered accumulation >1 quadrant and ≦3 quadrants; and grade 4, clustered accumulation ≧3
the change in minimum lumen area | 9 month
  absolute change in minimum lumen area between baseline and 36-week follow-up
the change in minimum lumen area | 9 month
  percentage of change in minimum lumen area between baseline and 36-week follow-up
the number of thin-cap fibroatheroma | 9 month
  change of the number of thin-cap fibroatheroma at 36-week follow-up
the change in total cholesterol | 9 month
  absolute change in serum level of of total cholesterol between baseline and 36-week follow-up
the change in total cholesterol | 9 month
  percent change in serum level of of total cholesterol between baseline and 36-week follow-up
the change in LDL-C | 9 month
  absolute change in serum level of of LDL-C between baseline and 36-week follow-up
the change in LDL-C | 9 month
  percentage change in serum level of of LDL-C between baseline and 36-week follow-up
the change in HDL-C | 9 month
  absolute change in serum level of of HDL-C between baseline and 36-week follow-up
the change in HDL-C | 9 month
  percentage change in serum level of of HDL-C between baseline and 36-week follow-up
the change in non-HDL-C | 9 month
  absolute change in serum level of of non-HDL-C between baseline and 36-week follow-up
the change in non-HDL-C | 9 month
  percentage change in serum level of of non-HDL-C between baseline and 36-week follow-up
the change in apolipoprotein B | 9 month
  absolute change in serum level of of apolipoprotein B between baseline and 36-week follow-up
the change in apolipoprotein B | 9 month
  percentage change in serum level of of apolipoprotein B between baseline and 36-week follow-up
the change in Lp(a) | 9 month
  absolute change in serum level of of Lp (a) between baseline and 36-week follow-up
the change in Lp(a) | 9 month
  percentage change in serum level of of Lp (a) between baseline and 36-week follow-up
the change in hs-CRP | 9 month
  absolute change in serum level of hs-CRP between baseline and 36-week follow-up
the change in hs-CRP | 9 month
  percentage change in serum level of hs-CRP between baseline and 36-week follow-up
the change in IL-1β | 9 month
  absolute change in serum level of IL-1β between baseline and 36-week follow-up
the change in IL-1β | 9 month
  percentage change in serum level of IL-1β between baseline and 36-week follow-up
the change in IL-6 | 9 month
  absolute change in serum level of IL-6 between baseline and 36-week follow-up
the change in IL-6 | 9 month
  percentage change in serum level of IL-6 between baseline and 36-week follow-up
the change in TNF-α | 9 month
  absolute change in serum level of TNF-α between baseline and 36-week follow-up
the change in TNF-α | 9 month
  percentage change in serum level of TNF-α between baseline and 36-week follow-up
the change in MCP-1 | 9 month
  absolute change in serum level of MCP-1 between baseline and 36-week follow-up
the change in MCP-1 | 9 month
  percentage change in serum level of MCP-1 between baseline and 36-week follow-up
the change in MMP-2 | 9 month
  absolute change in serum level ofMMP-2 between baseline and 36-week follow-up
the change in MMP-2 | 9 month
  percentage change in serum level ofMMP-2 between baseline and 36-week follow-up
the change in MMP-9 | 9 month
  absolute change in serum level of MMP-9 between baseline and 36-week follow-up
the change in MMP-9 | 9 month
  percentage change in serum level of MMP-9 between baseline and 36-week follow-up
the change in VCAM-1 | 9 month
  absolute change in serum level of VCAM-1between baseline and 36-week follow-up
the change in VCAM-1 | 9 month
  percentage change in serum level of VCAM-1 between baseline and 36-week follow-up
the change in ICAM-1 | 9 month
  absolute change in serum level of ICAM-1 between baseline and 36-week follow-up
the change in ICAM-1 | 9 month
  percentage change in serum level of ICAM-1 between baseline and 36-week follow-up
the change in free PCSK9 | 9 month
  absolute change in serum level of free PCSK9 between baseline and 36-week follow-up
the change in free PCSK9 | 9 month
  percentage change in serum level of free PCSK9 between baseline and 36-week follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Hiromasa Otake, M.D, Ph,D, Principal Investigator — Kobe University Graduate School of Medicine
Locations (1):
- Kobe University Graduate School of Medicine, Department of Cardiology, Kobe, Hyōgo, Japan

REFERENCES:
- [Derived] Otake H, Sugizaki Y, Toba T, Nagano Y, Tsukiyama Y, Yanaka KI, Yamamoto H, Nagasawa A, Onishi H, Takeshige R, Nakano S, Matsuoka Y, Tanimura K, Kawamori H, Shinke T, Hirata KI. Efficacy of alirocumab for reducing plaque vulnerability: Study protocol for ALTAIR, a randomized controlled trial in Japanese patients with coronary artery disease receiving rosuvastatin. J Cardiol. 2019 Mar;73(3):228-232. doi: 10.1016/j.jjcc.2018.11.012. Epub 2018 Dec 19. PMID 30579806